CLINICAL TRIAL: NCT01030666
Title: Effect of Postsurgical Systemic Doxycycline After Regenerative Periodontal Therapy. A Randomized Placebo-controlled Clinical Trial
Brief Title: Effect of Postsurgical Systemic Doxycycline After Regenerative Periodontal Therapy
Acronym: GTRDOXY
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: shelf life of investigational drug ran out before 90 patients could be included
Sponsor: Peter Eickholz (Other)
Collaborators: Heidelberg University (Other); Dr. August Wolff GmbH & Co. KG Arzneimittel (Industry); Gaba International AG (Industry)
Responsible Party: Sponsor-Investigator, Peter Eickholz, Prof. Dr. med. dent., Goethe University
Organization: Goethe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DoxP-01/2006
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Results first posted 2012-11-27 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-09

CONDITIONS: Periodontitis
Keywords: periodontal regeneration; radiographic bone fill; infrabony defects; randomized placebo-controlled clinical trial; guided tissue regeneration, periodontal
MeSH Terms: conditions — Periodontitis | interventions — Doxycycline; Tooth Exfoliation; enamel matrix proteins; Chlorhexidine; Ibuprofen; chlorhexidine gluconate; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- doxycycline (Experimental): The patients of the doxycycline group will take 200 mg doxycycline once a day for 7 days after regenerative therapy of an infrabony defects
  * modified/simplified papilla preservation flap; scaling
  * Prefgel/Emdogain
  * 0.12% chlorhexidine gluconate solution
  * Ibuprofen 400 mg (if necessary)
  * 1% chlorhexidine gluconate gel (if necessary)
  Interventions: Drug: Doxycycline; Procedure: modified/simplified papilla preservation flap; scaling; Biological: Prefgel/Emdogain; Drug: 0.12% chlorhexidine gluconate solution; Drug: Ibuprofen 400 mg (if necessary); Drug: 1% chlorhexidine gluconate gel (if necessary)
- placebo (Placebo Comparator): The patients of the control group will take placebo once a day for 7 days after regenerative therapy of an infrabony defect
  * modified/simplified papilla preservation flap; scaling
  * Prefgel/Emdogain
  * 0.12% chlorhexidine gluconate solution
  * Ibuprofen 400 mg (if necessary)
  * 1% chlorhexidine gluconate gel (if necessary)
  Interventions: Drug: Placebo; Procedure: modified/simplified papilla preservation flap; scaling; Biological: Prefgel/Emdogain; Drug: 0.12% chlorhexidine gluconate solution; Drug: Ibuprofen 400 mg (if necessary); Drug: 1% chlorhexidine gluconate gel (if necessary)

INTERVENTIONS:
Drug: Doxycycline — The patients of the doxycycline group will take 200 mg doxycycline once a day for 7 days after regenerative therapy of an infrabony defects.
  Other Names: Doxy-Wolff 200
  Arms: doxycycline
Drug: Placebo — The patients of the doxycycline group will take 200 mg placebo once a day for 7 days after regenerative therapy of an infrabony defects.
  Arms: placebo
Procedure: modified/simplified papilla preservation flap; scaling — Following an intra-crevicular incision a mucoperiosteal flap was reflected to a height of 5 mm exposing the bony margin of the defect and allowing complete visualization of the infrabony lesion. The flap was designed according to the modified or simplified papilla preservation technique to obtain primary closure of the wound and the membrane respectively. The flap was extended at least one tooth mesially and distally of the defect side. After complete removal of inflammatory granulation tissue, the root surfaces were thoroughly scaled and root planed.
Biological: Prefgel/Emdogain — When using EMD the root surfaces facing the infrabony defect were conditioned with EDTA (prefgel; Institut Straumann AG, Basel, Switzerland) for 2 min. first. Then the EDTA was washed out with plenty of saline. After drying the surfaces EMD was applied starting at the bottom of the defect and proceeding coronally.
  Other Names: EDTA/Enamel matrix derivative (EMD)
Drug: 0.12% chlorhexidine gluconate solution — Furthermore, all patients were advised to rinse with a 0.12% chlorhexidine gluconate solution (ParoEx; Butler, Kriftel, Germany) for 2 min. twice daily for 5-7 weeksafter surgery.
  Other Names: ParoEx
Drug: Ibuprofen 400 mg (if necessary) — 400 mg ibuprofen qd was prescribed for patient's comfort if necessary.
Drug: 1% chlorhexidine gluconate gel (if necessary) — If soft tissue dehiscence was noted the patient was advised to use a 1% chlorhexidine gluconate gel (Chlorhexamed 1% Gel; GlaxoSmithKline, Bühl, Germany) twice daily
  Other Names: Chlorhexamed 1% Gel

SUMMARY:
Study Hypothesis: The administration of 200 mg doxycycline once a day for 7 days after regenerative periodontal therapy of infrabony defects improves the results of therapy (clinical vertical attachment gains [CAL-V], bony fill) and reduces postoperative flap dehiscence and defect exposure.

In each of 90 patients one infrabony defect shall be treated by regenerative techniques (guided tissue regeneration [GTR], enamel matrix derivative [EMD]). Prior to , 6, 12, and 24 months after surgery clinical measurements (Plaque Index [PlI], probing depth [PD], vertical clinical attachment level [CAL-V], Gingival Index [GI]) and standardized radiographs are obtained.

DETAILED DESCRIPTION:
Patients From April 2007 until February 2009 all patients undergoing periodontal treatment at the Department of Periodontology, Center of Dental, Oral, and Maxillofacial Medicine (Carolinum), Johann Wolfgang Goethe-University Frankfurt/Main and the Section of Periodontology, Department of Conservative Dentistry, Clinic for Oral, Dental and Maxillofacial Diseases, University Hospital Heidelberg are screened for this study. Patients and methods of this study have been described in detail before. Thus only a brief description is provided.

The trial is approved by the Institutional Review Boards for Human Studies of the Medical Faculties of the Johann Wolfgang Goethe-University Frankfurt/Main (159/06) and the University of Heidelberg (ABmu-179/2006) as well as the German Federal Drug Authority (Bundesamt für Arzneimittel und Medizinprodukte). All participating individuals are informed on risks, benefit and the procedures of the study. All give written informed consent. The study is registered under the EudraCT-Nr. 2006-001367-36 and under the number NCT01030666.

Clinical measurements The following clinical parameters are assessed at six sites per tooth (mesiobuccal, midbuccal, distobuccal, distolingual, midlingual, mesiolingual) at baseline, 12, and 24 months after surgery: Gingival Index (GI), Plaque Index (PI), PD and CAL-V to the nearest 0.5 mm using a straight manual periodontal probe (PCPUNC 15, Hu Friedy, Chicago, IL, USA). As reference for the CAL-V measurements, the cemento-enamel junction (CEJ) is used. If the CEJ is destroyed by a restoration the restoration margin (RM) serves as reference.

Radiographic examination Standardized radiographs are obtained of test teeth by modified film holders (VIP 2 Positioning, UpRad Corp., Fort Lauderdale, FL, USA). These are done routinely in the clinical setting, after antiinfective and immediately before surgical treatment. Intraoral size 0 and 2 dental films (Insight, Eastman Kodak Co., Rochester, NY, USA) are exposed using an x-ray source (Heliodent DS, Sirona, Bensheim, Germany) with 7 mA and 60 kVp and developed under standardized conditions (XR24pro, Dürr Dental GmbH, Bietigheim-Bissingen, Germany).

Radiographic evaluation All radiographs are evaluated by one examiner (LR) who is blinded to the clinical results and to the time point the particular radiographs had been taken. All radiographs are digitalized using a computer program (SIDEXIS nextGeneration 1.51, Sirona, Bensheim, Germany) and a flatbed scanner (Microtek ScanMaker 4, Microtek, Hsinchu, Taiwan) with 600 dpi resolution and 8 bit grey values. The image files are stored as TIFF files and analyzed using the above mentioned computer program (SIDEXIS nextGeneration 1.51, Sirona, Bensheim, Germany) and a 19' flat Screen (Totoku CCL 192 plus, Totoku Electric, Ueda, Japan).

For evaluation the analyzing tool of the program (SIDEXIS nextGeneration 1.51, Sirona, Bensheim, Germany) is used. The image files are opened and magnified by using the function "zoom" once. Then the distances CEJ/RM to alveolar crest (AC), CEJ/RM to bony defect (DB), and the depth of the infrabony component (INFRA) are measured. The definition of these radiographic landmarks has been published in detail before.

Microbiological examination Immediately before and 14±2 days after surgery subgingival plaque samples are taken from the test sites of and analyzed by a commercially available real-time PCR test (Meridol Paro Diagnostik, GABA GmbH, Lörrach, Germany) for Aggregatibacter actinomycetemcomitans (A.a.), Porphyromonas gingivalis (P.g.), Tannerella forsythia (T.f.), Treponema denticola (T.d.), Fusobacterium nucleatum (F.n.), and Prevotella intermedia (P.i.). The detection limit of this test is 10².

Periodontal Surgery Infrabony defects reported in this analysis are treated by application of EMD (Emdogain®, Institut Straumann AG, Basel, Switzerland). Before closure of the defect intrasurgical parameters are measured.

Postsurgical Care

All patients take a postsurgical medication once a day for 7 days after regenerative periodontal therapy:

* Test: 200 mg doxycycline
* Control: 200 mg placebo. Doxycycline and placebo are packaged identically and stored in sealed envelopes that were marked with the randomization code. Patients receive doxycycline or placebo after regenerative surgery is accomplished. Patient and clinician are blinded. Block randomization by smoking status (current smoking: smokers/former and never smoking: non smokers) is provided by the manufacturer of the doxycycline (August Wolff GmbH & Co. Arzneimittel, Bielefeld, Germany).

Further, all patients are advised to rinse with a 0.12 % chlorhexidine gluconate solution (ParoEx, Butler, Kriftel, Germany) for 2 minutes bd for 5 to 7 weeks after surgery. During this time, all patients have to refrain from individual mechanical plaque control and thus are seen every other week for control and gentle cleaning of the teeth. In addition, 400 mg ibuprofen qd is prescribed for patient's comfort if necessary. If soft tissue dehiscence is noted the patient is advised to use a 1 % chlorhexidine gluconate gel (Chlorhexamed 1% Gel, GlaxoSmithKline, Bühl, Germany) twice daily. Sutures are retained as long as they maintained closure.18 Seven to 8 days after surgery wound healing is classified according to the Early Wound-Healing Index (EWI).

Statistical analysis Sample size calculation is based on an observed standard deviation for CAL-V gain (1.6 mm) in a study comparing regenerative therapy with and without antibiotics. To detect a mean difference of 1.0 mm with a test power of 80% and a type 1 error alpha < 0.05 a minimal sample size of 84 patients has to be recruited, 42 for each group. Thus, it is decided to recruit a total of 90 patients.

The patient is defined as statistical unit. CAL-V gain at 6 months is used as primary and bony fill at 12 months as secondary outcome variables. All other parameters are control variables. Baseline patient characteristics are described as means±SD (age, PCR) or frequencies/percentages (sex, smoking). All clinical parameters are calculated as means±SD (PI, GI, PD, CAL-V, INFRA).

After controlling for normal distribution CAL-V gain and PD reduction for the 2 test groups (DOXY/PLAC) are compared using an independent t test. Intragroup comparisons (baseline/12/24 months) are calculated using the paired t test. Inter and intragroup comparisons for radiographic bone, PI and GI are calculated using Mann Whitney U and Wilcoxon test, respectively. To explore the impact of subgingival microflora on the primary and secondary outcome variables we compare CAL-V gain (independent t test) 6 months and bony fill (Mann Whitney U) 12 months after therapy according to presence/absence of the tested periodontal pathogens.

A multiple regression model is calculated for the dependent variable bony fill with the independent variables baseline clinical parameters (CAL-V, PD, GI, PI), postsurgical medication (DOXY/PLAC), defect parameters (INFRA, % 1, 2, 3wall component), baseline A. actinomycetemcomitans, age, sex, centre, smoking, EHI. Sex, centre, and smoking habits are defined by indicator variables. All patients that are recruited and treated according to the study protocol are considered for analysis (intent to treat: ITT). If a patient left the study before finishing all re-examinations the respective data of the last re-examination are entered into the analysis (last observation carried forward: LOCF). Statistical analysis is performed using a PC program (SystatTM for Windows Version 10, Systat Inc. Evanston, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (at least 18 years of age) with moderate to severe periodontal disease (chronic and aggressive periodontitis) to be recruited from the Dept. of Periodontology, Centre for Dental, Oral, and Maxillofacial Medicine, Hospital of the Johann Wolfgang Goethe-University Frankfurt/Main and from the Section of Periodontology, Dept. of Conservative Dentistry, Clinic for Oral, Dental, and Maxillofacial Diseases, University Hospital Heidelberg
* completed initial periodontal treatment consisting of oral hygiene instruction, scaling and root planing under local anesthesia according the concept of full-mouth disinfection and re evaluation of the tissue response and the patient's plaque control 3 months later. Sites with infrabony defects and persisting pockets (PD > 5 mm and bleeding on probing, BOP) that occur at re evaluation or supportive periodontal treatment (SPT) are subjected to surgical therapy.
* at least one radiographically detectable infrabony lesion
* good physical health and with effective individual plaque control (Full-mouth-plaque score PCR </= 30% [O'Leary et al. 1972])
* interproximal angular defects on single-rooted teeth or multi-rooted teeth without furcation involvement, radiographic infrabony component >/= 4 mm, vertical clinical attachment loss (CAL-V) > 6 mm and PPD >/= 6 mm
* Only women in childbearing age (< 45 years) who provide contraception from screening to U2
* informed written consent

Exclusion Criteria:

* known allergies to tetracyclines or any components of the active drug or placebo
* severe liver dysfunction
* local or systemic antibiotic treatment during the last 3 months before surgery
* ineffective individual plaque control (PCR > 30%)
* kidney dysfunction
* medication with barbiturate, carbamazepin, diphenyhydantoine, sulfonyl-urea, methoxyflurane, ciclosporin A, theophylline, isotretionin
* chronic alcohol abuse
* anticoagulative therapy
* need for antibiotic endocarditis prophylaxis
* pregnancy
* lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-04; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Eickholz, Prof Dr, Principal Investigator — Dept. of Periodontology, Center for Dental, Oral, and Maxillofacial Medicine, Johann Wolfgang Goethe-University
Locations (2):
- Germany (2):
  - Dept. of Periodontology, Center of Dental, Oral, and Maxillofacial Medicine, Johann Wolfgang Goethe-University, Frankfurt am Main
  - Section of Periodontology, University Hospital Heidelberg, Heidelberg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rollke L, Schacher B, Wohlfeil M, Kim TS, Kaltschmitt J, Krieger J, Krigar DM, Reitmeir P, Eickholz P. Regenerative therapy of infrabony defects with or without systemic doxycycline. A randomized placebo-controlled trial. J Clin Periodontol. 2012 May;39(5):448-56. doi: 10.1111/j.1600-051X.2012.01861.x. Epub 2012 Mar 4. PMID 22385260
- [Result] Eickholz P, Rollke L, Schacher B, Wohlfeil M, Dannewitz B, Kaltschmitt J, Krieger JK, Krigar DM, Reitmeir P, Kim TS. Enamel matrix derivative in propylene glycol alginate for treatment of infrabony defects with or without systemic doxycycline: 12- and 24-month results. J Periodontol. 2014 May;85(5):669-75. doi: 10.1902/jop.2013.130290. Epub 2013 Sep 24. PMID 24059744

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From April 2007 to February 2009 all patients undergoing periodontal treatment at the Dept. of Periodontology, JWGUniversity Frankfurt and the Section of Periodontology, Department of Conservative Dentistry, University Hospital Heidelberg were screened for this study.
Groups:
- Placebo: The patients of the control group will take placebo once a day for 7 days after regenerative therapy of an infrabony defect
Period: Overall Study
Arm/Group | Doxycycline | Placebo
Started | 28 | 33
Completed | 25 | 31
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxycycline | Placebo | Total
Number analyzed (Participants) | 28 | 33 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 32 | 55
  >=65 years | 5 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (10.3) | 49.2 (10) | 51.5 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 23 | 34
  Male | 17 | 10 | 27
Region of Enrollment [Number; unit: participants]
  Germany | 28 | 33 | 61

OUTCOME MEASURES:

1. Primary Outcome: Vertical Clinical Attachment (PAL-V) Gain 6 Months After Surgery
Description: Difference of PAL-V measurement at baseline and 6 months. PAL-V were measured to the nearest 0.5 mm using a straight manual periodontal probe (PCPUNC 15, Hu Friedy, Chicago, IL, USA). As reference for the PAL-V measurements, the cemento-enamel junction (CEJ) was used. If the CEJ is destroyed by a restoration (filling, crown) the margin of this restoration served as reference.
Time Frame: Baseline to 6 months after surgery
Population: per protocol analysis: all participants who attended the 6 months re-examination
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Doxycycline: The patients of the doxycycline group will take 200 mg doxycycline once a day for 7 days after regenerative therapy of an infrabony defects addionally to
  * modified/simplified papilla preservation flap; scaling
  * Prefgel/Emdogain
  * 0.12% chlorhexidine gluconate solution
  * Ibuprofen 400 mg (if necessary)
  * 1% chlorhexidine gluconate gel (if necessary)
- Placebo: The patients of the control group will take placebo once a day for 7 days after regenerative therapy of an infrabony defect additionally to
  * modified/simplified papilla preservation flap; scaling
  * Prefgel/Emdogain
  * 0.12% chlorhexidine gluconate solution
  * Ibuprofen 400 mg (if necessary)
  * 1% chlorhexidine gluconate gel (if necessary)
Arm/Group | Doxycycline | Placebo
Number analyzed (Participants) | 27 | 31
mm | 3.11 (1.50) | 3.40 (1.79)

2. Secondary Outcome: Radiographic Bony Fill 12 Months After Surgery (Reduction of Distance Cemento-enamel Junction [CEJ] to Bony Defect [BD])
Description: If the CEJ was destroyed by the restorative treatment the margin of the restoration was taken as landmark. BD is defined as most coronal point where the periodontal ligament space shows a continuous width. If no periodontal ligament space could be identified, the point where the projection of the alveolar crest (AC) crossed the root surface was taken as a landmark. If both structures could be identified at one defect, the point defined by the periodontal ligament was used as BD and the crossing of the silhouette of the alveolar crest with the root surface was defined as AC. If several bony contours could be identified, the most apical one that crossed the root was defined as the BD and the most coronal one as AC.
Time Frame: Baseline to 12 months after surgery
Population: ITT population. Missing data due to losing to follow-up: last observation carried forward. Patients whose radiographs could not be analysed were excluded.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Doxycycline: The patients of the doxycycline group will take 200 mg doxycycline once a day for 7 days after regenerative therapy of an infrabony defects additionally to
  * modified/simplified papilla preservation flap; scaling
  * Prefgel/Emdogain
  * 0.12% chlorhexidine gluconate solution
  * Ibuprofen 400 mg (if necessary)
  * 1% chlorhexidine gluconate gel (if necessary)
Arm/Group | Doxycycline | Placebo
Number analyzed (Participants) | 25 | 30
mm | 1.09 (2.7) | 1.51 (2.89)

ADVERSE EVENTS:
Arm/Group | Doxycycline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/33
Other Adverse Events (participants affected / at risk) | 8/28 | 9/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxycycline (N=28) | Placebo (N=33)
head ache (Nervous system disorders) | 1 (1) | 4 (4)
Nausea (Ear and labyrinth disorders) | 3 (3) | 1 (1)
tiredness (General disorders) | 0 (0) | 2 (2)
tooth discomfort/pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
mucosal/skin lesions (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
The study had to be terminated due to shelf life of test drug running out prior to including 90 patients resulting in the low test power of 50%.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No